CLINICAL TRIAL: NCT02862587
Title: Clinical Study Using Precision Cell Immunotherapy Combined With Transcatheter Arterial Chemoembolization in Advanced Liver Cancer
Brief Title: Precision Cell Immunotherapy Combined With TACE in Advanced Liver Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai International Medical Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIMC-20160104
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Precision Cells; Chemotherapy; Advanced Lung Cancer
Keywords: Precision Cells; Chemotherapy; Advanced Lung Cancer
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Precision Cells (Experimental): precision cells combined with Chemotherapy treatment:
  Chemotherapy:
  once a week with a total of six times before 60 days prior to the start of drawing blood. precision cells：once per 3 weeks with a total of three periods.
  Interventions: Drug: Chemotherapy; Biological: precision cells
- Chemotherapy (Active Comparator): Once a week with a total of six times before 60 days prior to the start of drawing blood.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Cisplatin：60mg/m2，Gemcitabine：1g/m2,Physiological saline 100ml:IV (in the vein) once a week with a total of six times.
Biological: precision cells — precision cells DC cell suspension (1×10*7 DC+physiological saline + 0.25% human bloodalbumin)1ml for each infusion, subcutaneous injection for each infusion, 3 cycles, each cycle received two infusions on day 19, 20; 40, 41; 61, 62. PNAT/PMAT cell suspension (1-6×109 PNAT + physiological saline + 0.25% human bloodalbumin) 300ml for each infusion, IV (in the vein) for each infusion, 3 cycles, each cycle received one infusions on day 21, 42, 63.
  Arms: Precision Cells

SUMMARY:
Objectives:

To evaluate the safety and effectiveness of cell therapy using precision cells to treat Advanced Lung Cancer.

Eligibility:

Individuals greater than or equal to 18 years of age and less than or equal to 65 years of age who have been diagnosed with Advanced Lung Cancer.

DETAILED DESCRIPTION:
A total of 40 patients may be enrolled over a period of 1-2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 18~65 years old, male or female;
* Life expectancy≥6 months;
* ECOG score: 0-3;
* Advanced Malignancies (lung cancer) were diagnosed by pathological or clinical physicians;
* Enough venous channel, no other contraindications to the separation and collection of white blood cells;
* Laboratory examination: white blood cell≥3 x 10*9/L, blood platelet count≥60 x 10*/L,hemoglobin≥85g/L; lymphocyte count≥15%, total bilirubin≤100 mol/L; ALT and AST less than five times of the normal level; serum creatinine less than 1.5 times of the normal level;
* Signed informed consent;
* Women of child-bearing age must have evidence of negative pregnancy test and be willing to practice birth control after 2 weeks following the cells transfusion.

Exclusion Criteria:

* Expected Overall survival < 6 months;
* Patients with uncontrolled hypertension (>160/95mmHg), unstable coronary disease (uncontrolled arrhythmias, unstable angina, decompensated congestive heart failure (> Class II, NYHA), or myocardial infarction within 6 months;
* Other serious diseases: nervous, mental disorders, immune regulatory diseases, metabolic diseases, infectious diseases, etc;
* Other drugs, or other biological treatment,chemotherapy or radiotherapy are performed within a month;
* Unable or unwilling to provide informed consent, or fail to comply with the test requirements.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-03 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
Progress-free survival | 2 years

SECONDARY OUTCOMES:
Quality of life | 2 years
  Questionnaire will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai International Medical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No